CLINICAL TRIAL: NCT04114708
Title: MRI Review of ACLR With and Without Lateral Extra-articular Tenodesis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-01185
Record Dates: First submitted 2019-09-24; First posted 2019-10-03 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Ruptured Achilles Tendon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- ACLR (Other): All patients will undergo an anatomic ACLR via a standardized fashion using BTB autogaft graft.
  Interventions: Diagnostic Test: Anterior cruciate ligament Reconstruction (ACLR)
- ACLR with lateral extra-articular tenodesis (Other): All LETs will be performed in a standardized fashion using the modified Lameire technique.
  Interventions: Diagnostic Test: ACLR with lateral extra-articular tenodesis (LET)

INTERVENTIONS:
Diagnostic Test: Anterior cruciate ligament Reconstruction (ACLR) — All patients will undergo an anatomic ACLR via a standardized fashion using BTB autograft.
  Arms: ACLR
Diagnostic Test: ACLR with lateral extra-articular tenodesis (LET) — All LETs will be performed in a standardized fashion using the modified Lameire technique. All patients will undergo an anatomic ACLR via a standardized fashion using BTB autogaft graft.
  Arms: ACLR with lateral extra-articular tenodesis

SUMMARY:
The purpose of the proposed study is to evaluate the effect of lateral extra-articular tenodesis (LET) on anterior cruciate ligament reconstruction through evaluation of postoperative magnetic resonance imaging (MRI). This will be a single-center non-randomized controlled study. The study is comparing postoperative graft MRI findings in two cohorts: patients undergoing isolated ACLR and patients undergoing ACLR with lateral extra-articular tenodesis (LET). Postoperative MRIs will be obtained at 6, 9 and 12 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* ACL deficient knee
* skeletally mature (as defined by closed growth plates on plain radiograph)
* at least 13 years of age
* less than 26 years of age
* not pregnant
* two or more of following criteria: competitive pivoting sport, grade 2 pivot shift or - greater, generalized ligament laxity (beighton score of 4 or greater )
* no concomitant lateral meniscus tear

Exclusion Criteria:

* knee with intact ACL
* skeletally immature (as defined by open physis on plain radiograph)
* less than two of following criteria: competitive pivoting sport, grade 2 pivot shift or - greater, generalized ligament laxity (beighton score of 4 or greater )
* pregnant
* less than 13 years of age
* older than age 25
* previous ACL repair
* concomitant lateral meniscus tear
* unable to speak english or perform informed consent
* multiligamentous knee injury (two or more ligaments requiring surgical attention)
* varus or valgus malalignment greater than 3 degrees

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Determine if ACLR supplementation with LET results in superior MRI findings relative to ACLR alone | 1 Year
  MRI findings will be compared in patients receiving ACLR+LET versus just ACLR

SECONDARY OUTCOMES:
Graft Failure | 1 Year
  Defined as either symptomatic instability requiring revision or symptomatic instability with positive pivot shift or asymmetrical pivot shift greater than the contralateral side.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Alaia, MD, Principal Investigator — New York Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Requests should be directed to david.bloom@nyulangone.org To gain access, data requestors will need to sign a data access agreement.